CLINICAL TRIAL: NCT05825040
Title: Randomized Controlled Trial on Precision Mental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie W.S. MAK, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMHICS-HK
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Mental Well-being; Mental Health Issue; Mental Health Wellness 1; Precision Mental Health
Keywords: Online Psychological Intervention; Mental health; Mental well-being; Precision Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Online guided transdiagnostic cognitive behavioral therapy (Experimental): In the online guided transdiagnostic cognitive behavioral therapy group, participants will go through 8 modules with coach support in 8 weeks. They will complete 6 sets of questionnaires at the beginning of the study, at the 4th, 8th, and 16th weeks, and at 6 and 12 months after group allocation. All participants will be able to access all psychological interventions after they have completed the research.
  Interventions: Behavioral: Online guided transdiagnostic cognitive behavioural therapy
- Online self-guided transdiagnostic cognitive behavioral therapy (Experimental): In the online self-guided transdiagnostic cognitive behavioral therapy group, participants will go through 8 modules without coach support in 8 weeks. They will complete 6 sets of questionnaires at the beginning of the study, at the 4th, 8th, and 16th weeks, and at 6 and 12 months after group allocation. All participants will be able to access all psychological interventions after they have completed the research.
  Interventions: Behavioral: Online self-guided transdiagnostic cognitive behavioural therapy
- Waitlist control group (No Intervention): In the waitlist control group, participants are to refrain from using online psychological interventions until they finished the final questionnaire. They will complete 4 sets of questionnaires at the beginning of the study, at the 4th, 8th, and 16th weeks and at 6 and 12 months after group allocation. All participants will be able to access all psychological interventions after they have completed the research.
- Online self-guided mindfulness-based intervention (Experimental): In the online self-guided mindfulness-based intervention group, participants will go through 6 modules in 8 weeks without coach support. They will complete 6 sets of questionnaires at the beginning of the study, at the 4th, 8th, and 16th weeks, and at 6 and 12 months after group allocation. All participants will be able to access all psychological interventions after they have completed the research.
  Interventions: Behavioral: Online self-guided mindfulness-based intervention

INTERVENTIONS:
Behavioral: Online guided transdiagnostic cognitive behavioural therapy — The contents of guided transdiagnostic cognitive behavioural therapy are developed by clinical psychologists and psychological well-being officers. The intervention consists of 8 modules. Contents include emotional awareness, physical sensation, emotion-driven behavior, behavioral activation, worry, cognitive restructuring, behavioral experiment, and relapse prevention. Customized guidance will be provided by coaches once a week based on participants' performance
  Arms: Online guided transdiagnostic cognitive behavioral therapy
Behavioral: Online self-guided transdiagnostic cognitive behavioural therapy — The contents of self-guided transdiagnostic cognitive behavioural therapy are developed by clinical psychologists and psychological well-being officers. The intervention consists of 8 modules. Contents include emotional awareness, physical sensation, emotion-driven behavior, behavioral activation, worry, cognitive restructuring, behavioral experiment, and relapse prevention. No customized guidance will be provided to participants in the self-guided group.
  Arms: Online self-guided transdiagnostic cognitive behavioral therapy
Behavioral: Online self-guided mindfulness-based intervention — The contents of online self-guided mindfulness-based intervention are developed by clinical psychologists and psychological well-being officers. The intervention consists of 6 modules. Contents include mindfulness and auto-pilot, react and respond, aversion, craving, equanimity, and 'suffering', thoughts and letting go, starting with loving kindness, and mindfulness in life.
  Arms: Online self-guided mindfulness-based intervention

SUMMARY:
The current study aims to evaluate the effectiveness of different online psychological interventions, including guided and unguided transdiagnostic cognitive behavioural therapy, and unguided mindfulness-based intervention, on mental well-being in comparison to waitlist control. It is hypothesized that participants with the guided psychological intervention will show (H1) a greater reduction in mental health symptoms, and (H2) better mental well-being compared with participants with unguided psychological intervention and the control condition.

DETAILED DESCRIPTION:
In Hong Kong, insufficient resources in the current public health system lead to a long waiting time. Mental health services provided by the public health system mainly rely on traditional one-to-one face-to-face sessions. In the past 12 months, there were 47,879 new bookings in public psychiatry outpatient clinics and the longest waiting time was 94 weeks. Priority is always given to people with more severe mental health issues, which causes long waiting time for people with mild mental health symptoms. Untreated mental health issues can be escalated to more severe symptoms. Thus, in addition to treating mental illness, preventing common mental health issues and fostering mental health self-care in the general population are crucial to promote public mental health and reduce the illness burden in society.

Rather than resorting to mental health professionals for face-to-face service to treat common mental health concerns, digital technology provides a highly scalable and accessible means through which individuals can access mental health resources for self-care. Internet-delivered psychological therapy is one of the viable options for this situation. Internet-delivered cognitive behavioural therapy (ICBT) has been recommended by the NICE guidelines as one of the low-intensity interventions for people with depression and anxiety. Online scientific evidence-based psychological interventions provide solutions for the service users on their mental well-being issues without practical burdens resulted from long waiting time, high expenses, and stigmatization.

Internet-delivered mindfulness-based intervention (MBI) have emerged as a promising approach in reducing depressive and anxiety symptoms and improving mental well-being. A meta-analysis found that online MBIs had beneficial impact on depression, anxiety, well-being and mindfulness. It also found that guided online MBIs had larger effects on stress and mindfulness compared to unguided MBIs.

In this study, participants will be recruited through (1) advertising on online networking platforms (e.g., Facebook and Instagram), (2) mass mailing at investigator's institutions, and (3) snowball sampling.

Upon completing the screening and pre-evaluation questionnaire, participants will be randomly assigned to one of the groups based on computer-generated random digits. They will complete 5 more sets of questionnaires, including a mid-evaluation 4 weeks after group allocation, a post-evaluation 8 weeks after group allocation, and three follow-up questionnaires at 16 weeks, 6 months, and 12 months after group allocation. In experimental groups, participants will complete guided or self-guided transdiagnostic cognitive behavioural therapy, or self-guided mindfulness-based intervention within 8 weeks. In the waitlist control group, participants are to refrain from participating in psychological intervention until they finish the follow-up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 17 years old or above
* Able to read Chinese or English
* With internet connection and able to access the internet
* Does not register to Jockey Club TourHeart+ Project or participate in related research projects
* With moderate-severe GAD-7 a/o moderate-severe PHQ-9

Exclusion Criteria:

* People who are under 17 years old
* Cannot access the internet
* Existing users of Jockey Club TourHeart+ Project or participate in related research
* Without moderate-severe depressive or anxiety symptoms
* With suicidal risk

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire | 8th week
  It includes 9 items to assess the extent to which respondents are bothered by depression-related symptoms using a 4-point scale from 0 (not at all) to 3 (nearly every day). PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe levels of depression respectively (range: 0-27). PHQ-9 has sensitivity of 0.88 and specificity of 0.88 in detecting major depressive disorder (MDD) at a cut-off of 10. The internal consistency reliability of the Chinese version of the scale was 0.86.
Patient Health Questionnaire | 16th week
  It includes 9 items to assess the extent to which respondents are bothered by depression-related symptoms using a 4-point scale from 0 (not at all) to 3 (nearly every day). PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe levels of depression respectively (range: 0-27). PHQ-9 has sensitivity of 0.88 and specificity of 0.88 in detecting major depressive disorder (MDD) at a cut-off of 10. The internal consistency reliability of the Chinese version of the scale was 0.86.
Generalized Anxiety Disorder Assessment | 8th week
  It is a 7-item scale to assess the extent to which respondents are bothered by anxiety-related symptoms using a 4-point scale from 0 (not at all) to 3 (nearly every day). Scores of 5, 10, and 15 denote the mild, moderate, and severe levels of anxiety respectively (range: 0-21). At a cut-off of 10, GAD-7 has sensitivity of 0.89 and specificity of 0.82 in detecting generalized anxiety disorder (GAD). The internal consistency of the Chinese version was 0.93.
Generalized Anxiety Disorder Assessment | 16th week
  It is a 7-item scale to assess the extent to which respondents are bothered by anxiety-related symptoms using a 4-point scale from 0 (not at all) to 3 (nearly every day). Scores of 5, 10, and 15 denote the mild, moderate, and severe levels of anxiety respectively (range: 0-21). At a cut-off of 10, GAD-7 has sensitivity of 0.89 and specificity of 0.82 in detecting generalized anxiety disorder (GAD). The internal consistency of the Chinese version was 0.93.
The Short Warwick-Edinburgh Mental Wellbeing Scale | 8th week
  It contains 7 positively phrased items on a 5-point Likert scale from 1 (none of the time) to 5 (all of the time). Total scores ranged from 7 to 35, where higher scores indicated higher overall mental well-being. SWEMWBS satisfies the strict criteria for measurement demanded by the RASCH model and is preferable to the original 14-item WEMWBS scale. The Chinese version of SWEMWBS is reliable (Cronbach's alpha = 0.89) and has been validated among a sample in Hong Kong.
The Short Warwick-Edinburgh Mental Wellbeing Scale | 16th week
  It contains 7 positively phrased items on a 5-point Likert scale from 1 (none of the time) to 5 (all of the time). Total scores ranged from 7 to 35, where higher scores indicated higher overall mental well-being. SWEMWBS satisfies the strict criteria for measurement demanded by the RASCH model and is preferable to the original 14-item WEMWBS scale. The Chinese version of SWEMWBS is reliable (Cronbach's alpha = 0.89) and has been validated among a sample in Hong Kong.

SECONDARY OUTCOMES:
The Brief Experiential Avoidance Questionnaire (BEAQ) | 8th week
  The Brief Experiential Avoidance Questionnaire includes 15 items to measure experiential avoidance in 2 subscales: cognitive avoidance and behavioral avoidance. Items are rated on a 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). Item 6 is reverse-coded. The BEAQ shows good reliability (Cronbach's alpha = 0.80-0.89) for various samples.
The Brief Experiential Avoidance Questionnaire (BEAQ) | 16th week
  The Brief Experiential Avoidance Questionnaire includes 15 items to measure experiential avoidance in 2 subscales: cognitive avoidance and behavioral avoidance. Items are rated on a 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). Item 6 is reverse-coded. The BEAQ shows good reliability (Cronbach's alpha = 0.80-0.89) for various samples.
Behavioral Activation for Depression Scale - Short Form | 8th week
  The 9-item short version of Behavioral Activation for Depression Scale measures changes in activation and avoidance in the previous week. Items are rated on a 7-point Likert scale from 0 (not at all) to 6 (completely). Items 1, 6, 7, and 8 are reverse-coded. Higher scores on the total score represent increased activation. The BADS-SF has demonstrated good internal consistency (Cronbach's alpha = 0.82), construct validity, and predictive validity.
Behavioral Activation for Depression Scale - Short Form | 16th week
  The 9-item short version of Behavioral Activation for Depression Scale measures changes in activation and avoidance in the previous week. Items are rated on a 7-point Likert scale from 0 (not at all) to 6 (completely). Items 1, 6, 7, and 8 are reverse-coded. Higher scores on the total score represent increased activation. The BADS-SF has demonstrated good internal consistency (Cronbach's alpha = 0.82), construct validity, and predictive validity.
Intolerance of Uncertainty Scale (Short version) | 8th week
  The Intolerance of Uncertainty Scale - Short Version contains 12 items on a 5-point Likert scale from 1 (not at all characteristic of me) to 5 (entirely characteristic of me). It includes 2 subscales, prospective anxiety and inhibitory anxiety, which measure the approach-oriented and avoidance-oriented responses to uncertainty respectively. IUS-12 shows good reliability (Cronbach's alpha = 0.91) and convergent validity
Intolerance of Uncertainty Scale (Short version) | 16th week
  The Intolerance of Uncertainty Scale - Short Version contains 12 items on a 5-point Likert scale from 1 (not at all characteristic of me) to 5 (entirely characteristic of me). It includes 2 subscales, prospective anxiety and inhibitory anxiety, which measure the approach-oriented and avoidance-oriented responses to uncertainty respectively. IUS-12 shows good reliability (Cronbach's alpha = 0.91) and convergent validity
Emotion Regulation Questionnaire (ERQ) | 8th week
  It is a 10-item survey to assess two emotion-regulation strategies: cognitive reappraisal and expressive suppression. Items are rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). It demonstrated acceptable levels of reliability.
Emotion Regulation Questionnaire (ERQ) | 16th week
  It is a 10-item survey to assess two emotion-regulation strategies: cognitive reappraisal and expressive suppression. Items are rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). It demonstrated acceptable levels of reliability.
Anxiety Sensitivity Index-3 | 8th week
  It includes 18 items to measure the degree of physical, cognitive and social concerns about anxiety using a 5-point Likert scale from 0 (very little) to 4 (very much). ASI-3 is reliable (Cronbach's alpha = 0.79-0.91) with good convergent, discriminant and criterion-related validity and is preferable to the original ASI scale.
Anxiety Sensitivity Index-3 | 16th week
  It includes 18 items to measure the degree of physical, cognitive and social concerns about anxiety using a 5-point Likert scale from 0 (very little) to 4 (very much). ASI-3 is reliable (Cronbach's alpha = 0.79-0.91) with good convergent, discriminant and criterion-related validity and is preferable to the original ASI scale.
Ruminative response scale-short version | 8th week
  5 items from the brooding subscale are adopted to assess the passive thoughts to compare the current state with unrealistic standards using a 4-point Likert scale from 1 (almost never) to 4 (almost always). The brooding subscale demonstrated reliability (Cronbach's alpha = 0.77) and significant predictivity in depressive symptoms. The Chinese version of the scale was reliable and valid in examining rumination
Ruminative response scale-short version | 16th week
  5 items from the brooding subscale are adopted to assess the passive thoughts to compare the current state with unrealistic standards using a 4-point Likert scale from 1 (almost never) to 4 (almost always). The brooding subscale demonstrated reliability (Cronbach's alpha = 0.77) and significant predictivity in depressive symptoms. The Chinese version of the scale was reliable and valid in examining rumination
Nonattachment Scale-Short Form | 8th week
  Nonattachment Scale-Short Form (NAS-SF) includes 8 items to measure nonattachment using 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). It yielded satisfactory internal consistency and validity.
Nonattachment Scale-Short Form | 16th week
  Nonattachment Scale-Short Form (NAS-SF) includes 8 items to measure nonattachment using 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). It yielded satisfactory internal consistency and validity.
Need for autonomy | 8th week
  Two items adopted previous studies measure the need for autonomy. Items are rated on a 5-point Likert scale from 1 (completely disagree) to 5 (completely agree)
Patient Health Questionnaire | 6 months
  It includes 9 items to assess the extent to which respondents are bothered by depression-related symptoms using a 4-point scale from 0 (not at all) to 3 (nearly every day). PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe levels of depression respectively (range: 0-27). PHQ-9 has sensitivity of 0.88 and specificity of 0.88 in detecting major depressive disorder (MDD) at a cut-off of 10. The internal consistency reliability of the Chinese version of the scale was 0.86.
Patient Health Questionnaire | 12 months
  It includes 9 items to assess the extent to which respondents are bothered by depression-related symptoms using a 4-point scale from 0 (not at all) to 3 (nearly every day). PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe levels of depression respectively (range: 0-27). PHQ-9 has sensitivity of 0.88 and specificity of 0.88 in detecting major depressive disorder (MDD) at a cut-off of 10. The internal consistency reliability of the Chinese version of the scale was 0.86.
Generalized Anxiety Disorder Assessment | 6 months
  It is a 7-item scale to assess the extent to which respondents are bothered by anxiety-related symptoms using a 4-point scale from 0 (not at all) to 3 (nearly every day). Scores of 5, 10, and 15 denote the mild, moderate, and severe levels of anxiety respectively (range: 0-21). At a cut-off of 10, GAD-7 has sensitivity of 0.89 and specificity of 0.82 in detecting generalized anxiety disorder (GAD). The internal consistency of the Chinese version was 0.93.
Generalized Anxiety Disorder Assessment | 12 months
  It is a 7-item scale to assess the extent to which respondents are bothered by anxiety-related symptoms using a 4-point scale from 0 (not at all) to 3 (nearly every day). Scores of 5, 10, and 15 denote the mild, moderate, and severe levels of anxiety respectively (range: 0-21). At a cut-off of 10, GAD-7 has sensitivity of 0.89 and specificity of 0.82 in detecting generalized anxiety disorder (GAD). The internal consistency of the Chinese version was 0.93.
The Short Warwick-Edinburgh Mental Wellbeing Scale | 6 months
  It contains 7 positively phrased items on a 5-point Likert scale from 1 (none of the time) to 5 (all of the time). Total scores ranged from 7 to 35, where higher scores indicated higher overall mental well-being. SWEMWBS satisfies the strict criteria for measurement demanded by the RASCH model and is preferable to the original 14-item WEMWBS scale. The Chinese version of SWEMWBS is reliable (Cronbach's alpha = 0.89) and has been validated among a sample in Hong Kong.
The Short Warwick-Edinburgh Mental Wellbeing Scale | 12 months
  It contains 7 positively phrased items on a 5-point Likert scale from 1 (none of the time) to 5 (all of the time). Total scores ranged from 7 to 35, where higher scores indicated higher overall mental well-being. SWEMWBS satisfies the strict criteria for measurement demanded by the RASCH model and is preferable to the original 14-item WEMWBS scale. The Chinese version of SWEMWBS is reliable (Cronbach's alpha = 0.89) and has been validated among a sample in Hong Kong.
The Five Facet Mindfulness Questionnaire | 8th week
  It includes 20 items to measure mindfulness in 5 subscales: observing, describing, acting with awareness, nonjudging, and nonreacting. Items are rated on a 5-point scale from 1 (never or very rarely true) to 5 (very often true or always true). The FFMQ-C shows good test-retest reliability (0.88) and high internal consistency (Cronbach's alpha = 0.80-0,83) for various samples.
The Five Facet Mindfulness Questionnaire | 16th week
  It includes 20 items to measure mindfulness in 5 subscales: observing, describing, acting with awareness, nonjudging, and nonreacting. Items are rated on a 5-point scale from 1 (never or very rarely true) to 5 (very often true or always true). The FFMQ-C shows good test-retest reliability (0.88) and high internal consistency (Cronbach's alpha = 0.80-0,83) for various samples.

CONTACTS AND LOCATIONS:
Overall Officials: Winnie WS Mak, Principal Investigator — Professor
Locations (1):
- Diversity and Well-being Lab, Dept of Psychology, CUHK, Shatin, N.T., Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abd-Alrazaq AA, Alajlani M, Alalwan AA, Bewick BM, Gardner P, Househ M. An overview of the features of chatbots in mental health: A scoping review. Int J Med Inform. 2019 Dec;132:103978. doi: 10.1016/j.ijmedinf.2019.103978. Epub 2019 Sep 25. PMID 31622850
- [Background] Carleton RN, Norton MA, Asmundson GJ. Fearing the unknown: a short version of the Intolerance of Uncertainty Scale. J Anxiety Disord. 2007;21(1):105-17. doi: 10.1016/j.janxdis.2006.03.014. Epub 2006 May 2. PMID 16647833
- [Background] Chio, F. H., Lai, M. H., & Mak, W. W. (2018). Development of the Nonattachment Scale-Short Form (NAS-SF) using item response theory. Mindfulness, 9, 1299-1308.
- [Background] Choi I, Andrews G, Sharpe L, Hunt C. Help-seeking characteristics of Chinese- and English-speaking Australians accessing Internet-delivered cognitive behavioural therapy for depression. Soc Psychiatry Psychiatr Epidemiol. 2015 Jan;50(1):89-97. doi: 10.1007/s00127-014-0956-3. Epub 2014 Sep 6. PMID 25193374
- [Background] Dorow M, Lobner M, Pabst A, Stein J, Riedel-Heller SG. Preferences for Depression Treatment Including Internet-Based Interventions: Results From a Large Sample of Primary Care Patients. Front Psychiatry. 2018 May 17;9:181. doi: 10.3389/fpsyt.2018.00181. eCollection 2018. PMID 29867605
- [Background] Gamez W, Chmielewski M, Kotov R, Ruggero C, Suzuki N, Watson D. The brief experiential avoidance questionnaire: development and initial validation. Psychol Assess. 2014 Mar;26(1):35-45. doi: 10.1037/a0034473. Epub 2013 Sep 23. PMID 24059474
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] He J, Liu Y, Cheng C, Fang S, Wang X, Yao S. Psychometric Properties of the Chinese Version of the 10-Item Ruminative Response Scale Among Undergraduates and Depressive Patients. Front Psychiatry. 2021 May 26;12:626859. doi: 10.3389/fpsyt.2021.626859. eCollection 2021. PMID 34122165
- [Background] Hospital Authority. (n.d.). Waiting time for new case booking at Psychiatry specialist out-patient clinics. Retrieved March 20, 2022, from https://www.ha.org.hk/visitor/sopc_waiting_time.asp?id=7&lang=ENG
- [Background] Lam LC, Wong CS, Wang MJ, Chan WC, Chen EY, Ng RM, Hung SF, Cheung EF, Sham PC, Chiu HF, Lam M, Chang WC, Lee EH, Chiang TP, Lau JT, van Os J, Lewis G, Bebbington P. Prevalence, psychosocial correlates and service utilization of depressive and anxiety disorders in Hong Kong: the Hong Kong Mental Morbidity Survey (HKMMS). Soc Psychiatry Psychiatr Epidemiol. 2015 Sep;50(9):1379-88. doi: 10.1007/s00127-015-1014-5. Epub 2015 Feb 8. PMID 25660760
- [Background] Mak WW, Chan AT, Cheung EY, Lin CL, Ngai KC. Enhancing Web-based mindfulness training for mental health promotion with the health action process approach: randomized controlled trial. J Med Internet Res. 2015 Jan 19;17(1):e8. doi: 10.2196/jmir.3746. PMID 25599904
- [Background] Mak WW, Chio FH, Chan AT, Lui WW, Wu EK. The Efficacy of Internet-Based Mindfulness Training and Cognitive-Behavioral Training With Telephone Support in the Enhancement of Mental Health Among College Students and Young Working Adults: Randomized Controlled Trial. J Med Internet Res. 2017 Mar 22;19(3):e84. doi: 10.2196/jmir.6737. PMID 28330831
- [Background] Mak WW, Tong AC, Yip SY, Lui WW, Chio FH, Chan AT, Wong CC. Efficacy and Moderation of Mobile App-Based Programs for Mindfulness-Based Training, Self-Compassion Training, and Cognitive Behavioral Psychoeducation on Mental Health: Randomized Controlled Noninferiority Trial. JMIR Ment Health. 2018 Oct 11;5(4):e60. doi: 10.2196/mental.8597. PMID 30309837
- [Background] Manos RC, Kanter JW, Luo W. The behavioral activation for depression scale-short form: development and validation. Behav Ther. 2011 Dec;42(4):726-39. doi: 10.1016/j.beth.2011.04.004. Epub 2011 Jun 1. PMID 22036000
- [Background] NICE Guidance. (2018). Common mental health problems: Identification and pathways to care. Retrieved from https://www.nice.org.uk/guidance/cg123/resources/common-mental-health-problems-identification-and-pathways-to-care-pdf-35109448223173
- [Background] Ng SS, Lo AW, Leung TK, Chan FS, Wong AT, Lam RW, Tsang DK. Translation and validation of the Chinese version of the short Warwick-Edinburgh Mental Well-being Scale for patients with mental illness in Hong Kong. East Asian Arch Psychiatry. 2014 Mar;24(1):3-9. PMID 24676481
- [Background] Resnicow K, Zhou Y, Hawley S, Jimbo M, Ruffin MT, Davis RE, Shires D, Lafata JE. Communication preference moderates the effect of a tailored intervention to increase colorectal cancer screening among African Americans. Patient Educ Couns. 2014 Dec;97(3):370-5. doi: 10.1016/j.pec.2014.08.013. Epub 2014 Sep 3. PMID 25224317
- [Background] Schoofs, H., Hermans, D., & Raes, F. (2010). Brooding and reflection as subtypes of rumination: Evidence from confirmatory factor analysis in nonclinical samples using the Dutch Ruminative Response Scale. Journal of Psychopathology and Behavioral Assessment, 32, 609-617.
- [Background] Shek DTL, Dou D, Zhu X. Prevalence and Correlates of Mental Health of University Students in Hong Kong: What Happened One Year After the Occurrence of COVID-19? Front Public Health. 2022 Jun 29;10:857147. doi: 10.3389/fpubh.2022.857147. eCollection 2022. PMID 35844893
- [Background] Smit ES, Zeidler C, Resnicow K, de Vries H. Identifying the Most Autonomy-Supportive Message Frame in Digital Health Communication: A 2x2 Between-Subjects Experiment. J Med Internet Res. 2019 Oct 30;21(10):e14074. doi: 10.2196/14074. PMID 31670693
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Sun Y, Luk TT, Wang MP, Shen C, Ho SY, Viswanath K, Chan SSC, Lam TH. The reliability and validity of the Chinese Short Warwick-Edinburgh Mental Well-being Scale in the general population of Hong Kong. Qual Life Res. 2019 Oct;28(10):2813-2820. doi: 10.1007/s11136-019-02218-5. Epub 2019 May 29. PMID 31144205
- [Background] Taylor S, Zvolensky MJ, Cox BJ, Deacon B, Heimberg RG, Ledley DR, Abramowitz JS, Holaway RM, Sandin B, Stewart SH, Coles M, Eng W, Daly ES, Arrindell WA, Bouvard M, Cardenas SJ. Robust dimensions of anxiety sensitivity: development and initial validation of the Anxiety Sensitivity Index-3. Psychol Assess. 2007 Jun;19(2):176-88. doi: 10.1037/1040-3590.19.2.176. PMID 17563199
- [Background] Treynor, W., Gonzalez, R., & Nolen-Hoeksema, S. (2003). Rumination reconsidered: A psychometric analysis. Cognitive therapy and research, 27, 247-259.
- [Background] Hou J, Wong SY, Lo HH, Mak WW, Ma HS. Validation of a Chinese version of the Five Facet Mindfulness Questionnaire in Hong Kong and development of a short form. Assessment. 2014 Jun;21(3):363-71. doi: 10.1177/1073191113485121. Epub 2013 Apr 16. PMID 23596271
- [Background] Spijkerman MP, Pots WT, Bohlmeijer ET. Effectiveness of online mindfulness-based interventions in improving mental health: A review and meta-analysis of randomised controlled trials. Clin Psychol Rev. 2016 Apr;45:102-14. doi: 10.1016/j.cpr.2016.03.009. Epub 2016 Apr 1. PMID 27111302